CLINICAL TRIAL: NCT01855971
Title: Estrogen Receptors Beta (ER-B) as Therapeutic Targets for the Improvement of Cognitive Performance in Fragile-X (TESXF)
Brief Title: "Using Epigallocatechin Gallate (EGCG) and Cognitive Training to Modulate Cognitive Performance in Patients With Fragile X Syndrome" (TESFX)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Rafael de la Torre, Pharm D, PhD, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TESXF
Record Dates: First submitted 2013-05-09; First posted 2013-05-17 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Fragile X Syndrome
MeSH Terms: conditions — Fragile X Syndrome | interventions — epigallocatechin gallate; Cognitive Training

STUDY DESIGN:
Intervention Model Description: The study lasts 7 months :
  * from day 0 to month 1, patients will receive placebo, in order to avoid the placebo effect of the treatment.
  * from month 1 to month 4 : patients will be divided in two cohorts, one group receiving ECGC (experimental group), and the other placebo (control group).
  * from mont 4 to month 7 : no treatment in given, only effects of cessation of treatment are observed.
  Patients from both arms will receive Cognitive training.
Who Masked: Participant, Investigator
Masking Description: Placebo medication consists in rice flour tablets, given to patients of control group with the same posology than the ones of the experimental group (2*200mg / day).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fragile X syndrome experimental group (Active Comparator): 1. Administration of 400 mg/day of epigallocatechin-3-gallate (EGCG). Life Extension, Mega Green Tea Extract Decaffeinated, a dietary supplement containing EGCG extract (45% EGCGC).
     Dosage form: capsules of 200mg Route of administration: orally Dosage: 2 capsules per day (400 mg EGCG/day) Frequency: one capsule in the morning (fasting state) and a second capsule in the afternoon (before dinner).
     Treatment period: 3 months (from month 1 to month 4)
  2. Cognitive training: non-pharmacological cognitive training 3 sessions per week (1 hour per session) by using the Feskits program.
  Interventions: Dietary Supplement: EGCG; Other: Cognitive training
- Fragile X syndrome control group (Placebo Comparator): 1. Placebo administration. Placebo consists in capsules containing rice flour. Dosage form: capsules Route of administration: orally Dosage: 2 capsules per day Frequency: one capsule in the morning (fasting state) and a second capsule in the afternoon (before dinner).
  2. Cognitive training: non-pharmacological cognitive training 3 sessions per week (1 hour per session) by using the Feskits program.
  Interventions: Dietary Supplement: Placebo; Other: Cognitive training

INTERVENTIONS:
Dietary Supplement: EGCG — Life Extension, Mega Green Tea Extract Decaffeinated is a dietary supplement containing EGCG extract (45% EGCG). This extract contains 98% total polyphenols and 45% epigallocatechin-3-gallate (EGCG). EGCG administration in Down syndrome patients will result in an improvement of their cognitive performance.
  Other Names: Epigallocatechin-3-gallate (EGCG)
  Arms: Fragile X syndrome experimental group
Dietary Supplement: Placebo — Same capsules containing rice flour. No active treatment is given.
  Other Names: Matched placebo
  Arms: Fragile X syndrome control group
Other: Cognitive training — Feskits program 3 times per week (1 hour/session) Patients in this arm of the trial carried out computerized online training drawn from the Feskits program (www.feskits.com), chosen to have attention, memory and executive function components. Specifically the sessions included the following exercises: sustained attention, attention/perception, working memory, auditory and visual memory, executive function and language.

SUMMARY:
Fragile X syndrome (FXS) presents alterations in synaptic plasticity that produce intellectual disability. can produce improvement. Estrogens (targeting Estrogen Receptors beta (ER-β) can act as neuroprotective agents, promoting synaptic plasticity and neurite outgrowth, and health benefits derived from flavonoids, as the flavonol epigallocatechin gallate (EGCG), phytoestrogens of natural origin are partially explained by their interaction with membrane ER. Selective ER-β flavonoids are thus good candidates for their therapeutic evaluation in intellectual disabilities. EGCG also targets central intracellular transduction signals altered in FXS and improves memory recognition in a FXS animal model(adenosine triphosphate (ATP)-inhibitor of phosphatidylinositol 3-kinase (PI3K)and mammalian target of rapamycin (mTOR) and extracellular signal-regulated kinase (ERK1/2). This study targets the synaptic plasticity alterations that underlie the learning and memory impairment but also the computational disability in FXS. The hypothesis is that EGCG can act by favoring the physiological processes involved in cognition.

ELIGIBILITY:
Inclusion Criteria:

* Molecular diagnosis of Fragile X syndrome (FXS)
* Males and females aged 12 to 60 years.
* Study participants must understand and accept experimental procedures and assent to participate in the study signing an informed consent.
* Parents or caregivers have to understand and accept experimental procedures and sign informed consent form.
* Use of effective contraceptive methods in female participants
* Regular menstrual cycle (26-32 days duration) in female subjects
* Moderate mental disability (IQ>40)
* Body mass index (BMI) comprised between 18.5 and 29.9 kg/m2, and body weight between 50 and 100 kg.
* Non-smokers
* Electroencephalogram record and general blood and urine analysis performed at screening visit should be within normal values. Minor or occasional variations in normal values are allowed if, in the opinion of Principal Investigator, taking into account the state of the science, they are not clinically significant, they do not pose risk for the subjects and they do not interfere in the evaluation of the investigational product. These variations and their non-relevance should be justified by writing.

Exclusion Criteria:

* Not fulfil inclusion criteria.
* Subjects with neurological disease other than FXS, relevant medical disease, co-morbid mental disorder or currently taking any treatment that could interfere with cognitive function or alter any key biomarkers and biochemical parameters analyzed.
* Having suffered from any major illness or undergoing major surgery in the last 12 months preceding the study.
* Regular ingestion of psychotropic drugs in the three months preceding the study. Exceptions were made for single doses of symptomatic medication administered up to the week preceding the trial.
* Current ingestion of vitamin supplements or catechins or non steroidal antiinflammatory drug (NSAID) in the two weeks preceding the study.
* History or clinical proof of gastrointestinal, hepatic or renal problems or any other cause that may alter processes of absorption, distribution, metabolism, or excretion of the drug, or that might suggest gastrointestinal irritation to drug.
* Subjects following a cognitive training.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2013-06-11 (Actual); Primary Completion 2015-07-31 (Actual); Study Completion 2015-10-31 (Actual)

PRIMARY OUTCOMES:
Change in Prepulse inhibition of acoustic startle response (PPI) | From presdose baseline to 3 and 6 months (after treatment)
  Neurophysiology exploration (electroencephalogram)
The Kaufman Brief Intelligence Test (K-BIT) | at screening
  Evaluates the intellectual status and significantly correlates with the WISC-III.The intellectual quotient (IQ) will correspond to the K-BIT standardized total score, which can range from 40 (very low) to 160 (very high).
Changes in psicomotor speed (Motor Screening test (MOT, CANTAB)) | From presdose baseline to 3 and 6 months (after treatment)
  To assess psychomotor speed and accuracy. Participants were instructed to touch a series of crosses that appeared randomly on the screen. Response latency (in milliseconds) (MOT: Mean latency [ms]) will be considered in the present study.
Changes in Simple Reaction Time (SRT; CANTAB) | From presdose baseline to 3 and 6 months (after treatment)
  explores general alertness and motor speed. Subjects had to press the button on a press pad every time a square appeared in the middle of the screen. Intervals between the examinee's response and the next stimulus were variable during the task.
Changes in Digit Span: forward and backward recall (WAIS-III) | From presdose baseline to 3 and 6 months (after treatment)
  Forward recall score provides a good measure of verbal attention and working memory span. Backward recall score is predominantly a measure of verbal working memory span. Subjects were required to listen to a series of numbers with randomized presentation, and then repeat them back. The length of the series increased upon the subject's success.
Changes in Spatial Span (SSP): forward and backward recall (CANTAB) | From presdose baseline to 3 and 6 months (after treatment)
  Forward recall is predominantly a measure of visual attention and memory span. Participants were shown a sequence of squares that turned into a different color, one at each time, in a specific temporal order and spatial location. The examinee had to reproduce the sequence by touching on the screen the squares in the same order as they were presented. The length of the sequence increases in accordance to the subject's correct answers. Participants were shown a sequence of squares that turned into a different color, one at each time, in a specific temporal order and spatial location. The examinee had to reproduce the sequence by touching on the screen the squares in the same order as they were presented. The length of the sequence increases in accordance to the subject's correct answers.
Changes in executive function (Word fluency test) | From presdose baseline to 3 and 6 months (after treatment)
  Subjects were asked to generate as many words as possible in 1 minute belonging to the specified category of "animals" (open ranged: 0 to n1). High scores (number of words) (Semantic Word Fluency) indicate greater verbal fluency ability.
Changes in in executive function (Tower of London-Drexel University (ToLDx)) | From presdose baseline to 3 and 6 months (after treatment)
  This test requires moving three different colored balls across three different sized pegs in order to replicate a goal configuration. Movements follow strict rules. Two training tasks were followed by 10 problems of increasing complexity. The task finalized after the examinee failed to solve two consecutive problems.
Changes in in executive function (Weigl Color-Form Sort Test) | From presdose baseline to 3 and 6 months (after treatment)
  This is a set-shifting task that assesses the ability to categorize across two dimensions: color and shape. Instructions for administration and scoring were taken from Strauss & Lewin. Test material consisted of 12 tokens: four circles, four triangles, and four squares, and shapes were colored blue, red, yellow or green. The 12 tokens were displayed unsorted in front of the examinee. In the first trial the examinee is required to sort the tokens in a way that they go together (color or shape).
Changes in executive function (Cats & Dogs Test) | From presdose baseline to 3 and 6 months (after treatment)
  This is a Stroop-like task assessing response inhibition, based on the original Day-Night task. In this test, a sequence of 16 pictures, 8 cats and 8 dogs arranged in a prefixed order, are presented to the examinee on a single strip of card. The task consists of two trials with two different conditions: a control trial and an experimental-inhibition trial.
Changes in memory and learning (Paired Associates Learning (PAL, CANTAB)) | From presdose baseline to 3 and 6 months (after treatment)
  In this task the participants are required to learn associations between an abstract visual pattern and its location. Each participant is presented with a number of white boxes, arranged in a circle around an empty central space in the screen. Each box "opens" to reveal what is underneath (empty, or with a unique abstract pattern) in a randomized order until the participant has revealed all the contents. Next, a single pattern is presented in the center of the screen and the subject is instructed to touch the box where that pattern has been shown during the presentation phase of the trial. The task increases in difficulty from 1 to 8 patterns.
Changes in memory and learning (Pattern Recognition Memory (PRM, CANTAB)) | From presdose baseline to 3 and 6 months (after treatment)
  Participants are presented with a series of two blocks of 12 abstract visual patterns that appear sequentially in the center of the computer screen. Patterns are designed so that they cannot easily be given verbal labels. Each pattern is shown for 3 seconds. In each of the 12 recognition trials, two patterns are presented: one familiar (from the series that the participants have already seen) and one novel pattern. The participant have to recognize the previously seen pattern. The same procedure is repeated with a second block of 12 new patterns but this time the recognition trial started 20 minutes after the presentation of this second block to provide a measure of delayed recall.
Changes in memory and learning (Cued Recall Test) | From presdose baseline to 3 and 6 months (after treatment)
  The test consisted of a list of 12 items, which have to be verbally recalled by the examinee during 3 trials of free and cued recall. The test start with a learning phase where the examinee is required to learn the list of 12 items using 12 images. Four pictures are presented at a time, one in each quadrant of a card. First, the examinee have to name each of the four pictures in the card, and secondly assign each picture according to a verbal category-cue given by the examiner.
Changes in language (Boston Naming Test ) | From presdose baseline to 3 and 6 months (after treatment)
  The test consists of 60 black and white pictures graded in naming difficulty. Each picture is presented individually. The examinee is asked to name each item, and when unable to do so spontaneously, the examiner provides semantic and/or phonemic cues.
Changes in language (Token Test ) | From presdose baseline to 3 and 6 months (after treatment)
  Test materials consists of 20 tokens in two shapes (circles and rectangles), two sizes (big and small), and five colors (red, black, yellow, white, and green). The tokens are laid out according to a fixed configuration in front of the examinee. The test requires the examinee to touch the tokens according to the oral commands provided by the examiner. Thirty-six commands are divided into six stages of increasing complexity.
Changes in Adaptive Behavior in daily living | From presdose baseline to 3 and 6 months (after treatment)
  ABAS-II is designed, according to AAMS guidelines, for evaluating adaptive skills in people with mental disabilities of a wide age range and across multiple environments. The ABAS-II tool for adults (ages 16 to 89) includes 5 subscales which assesses the individual's competence (in terms of behavior frequency) in 10 different skill áreas.
Changes in Quality of life (Kidscreen-27 (parents version)) | From presdose baseline to 3 and 6 months (after treatment)
  This instrument assesses quality of life from the child and adolescent's perspective in terms of their physical, mental, and social well-being, higher scores corresponding to a greater quality of life. The questionnaire measures five dimensions.
change sin quality of sleep (the Pittsburgh Sleep Quality Index (PSQI)) | From presdose baseline to 3 and 6 months (after treatment)
  This questionnaire evaluates the quality and patterns of sleep in older adults. It assesses sleep performance over the previous month across seven different domains: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Parents will self-report all answers to each of the seven areas.
Changes in disrupting behavior (the Aberrant Behavior Checklist (ABC-C)) | From presdose baseline to 3 and 6 months (after treatment)
  The ABC-C is a 58-item questionnaire for caregivers designed to assess the presence and severity of psychiatric symptoms and behavioral disturbance commonly exhibited by individuals with IDD. The questionnaire explores problem behaviors across 5 domains.

SECONDARY OUTCOMES:
Changes in Phosphatidylinositol 3-kinase/mammalian target of rapamycin (PI3K/mTOR) concentration | From presdose baseline to 3 and 6 months (after treatment)
  Concentrations of PI3K/mTOR in human lymphocites.
Changes in Lipid Oxidation Biomarkers | From presdose baseline to 3 and 6 months (after treatment)
  Concentrations in plasma of oxidized- LDL.
Changes in body analysis composition | From presdose baseline to 3 and 6 months (after treatment)
  Bioimpedance body analysis composition (TANITA)
changes in clinical chemistry biomarkers | From presdose baseline to 3 and 6 months (after treatment)
changes in hematology biomarkers | From presdose baseline to 3 and 6 months (after treatment)
changes in coagulation biomarkers | From presdose baseline to 3 and 6 months (after treatment)
changes in urine analysis | From presdose baseline to 3 and 6 months (after treatment)
Changes in extracellular signal-regulated kinase 1 (ERK) biomarker | From baseline to 7 months
  Concentrations of Kinase 1(ERK) activity in human lymphocytes.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael de la Torre, PhamD, Principal Investigator — Parc de Salut Mar
Locations (1):
- Parc de Salut MAR, Hospital del Mar Medical Research Institute-IMIM, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adachi N, Tomonaga S, Tachibana T, Denbow DM, Furuse M. (-)-Epigallocatechin gallate attenuates acute stress responses through GABAergic system in the brain. Eur J Pharmacol. 2006 Feb 15;531(1-3):171-5. doi: 10.1016/j.ejphar.2005.12.024. Epub 2006 Feb 2. PMID 16457806
- [Background] Berry-Kravis E, Knox A, Hervey C. Targeted treatments for fragile X syndrome. J Neurodev Disord. 2011 Sep;3(3):193-210. doi: 10.1007/s11689-011-9074-7. Epub 2011 Feb 19. PMID 21484200
- [Background] Campbell EL, Chebib M, Johnston GA. The dietary flavonoids apigenin and (-)-epigallocatechin gallate enhance the positive modulation by diazepam of the activation by GABA of recombinant GABA(A) receptors. Biochem Pharmacol. 2004 Oct 15;68(8):1631-8. doi: 10.1016/j.bcp.2004.07.022. PMID 15451406
- [Background] Gross C, Berry-Kravis EM, Bassell GJ. Therapeutic strategies in fragile X syndrome: dysregulated mGluR signaling and beyond. Neuropsychopharmacology. 2012 Jan;37(1):178-95. doi: 10.1038/npp.2011.137. Epub 2011 Jul 27. PMID 21796106
- [Background] Levenga J, de Vrij FM, Oostra BA, Willemsen R. Potential therapeutic interventions for fragile X syndrome. Trends Mol Med. 2010 Nov;16(11):516-27. doi: 10.1016/j.molmed.2010.08.005. Epub 2010 Sep 21. PMID 20864408
- [Background] Van Aller GS, Carson JD, Tang W, Peng H, Zhao L, Copeland RA, Tummino PJ, Luo L. Epigallocatechin gallate (EGCG), a major component of green tea, is a dual phosphoinositide-3-kinase/mTOR inhibitor. Biochem Biophys Res Commun. 2011 Mar 11;406(2):194-9. doi: 10.1016/j.bbrc.2011.02.010. Epub 2011 Feb 15. PMID 21300025
- [Background] Verkerk AJ, Pieretti M, Sutcliffe JS, Fu YH, Kuhl DP, Pizzuti A, Reiner O, Richards S, Victoria MF, Zhang FP, et al. Identification of a gene (FMR-1) containing a CGG repeat coincident with a breakpoint cluster region exhibiting length variation in fragile X syndrome. Cell. 1991 May 31;65(5):905-14. doi: 10.1016/0092-8674(91)90397-h. PMID 1710175
- [Background] Vignes M, Maurice T, Lante F, Nedjar M, Thethi K, Guiramand J, Recasens M. Anxiolytic properties of green tea polyphenol (-)-epigallocatechin gallate (EGCG). Brain Res. 2006 Sep 19;1110(1):102-15. doi: 10.1016/j.brainres.2006.06.062. Epub 2006 Jul 21. PMID 16859659
- [Background] Yang J, Han Y, Sun H, Chen C, He D, Guo J, Yu C, Jiang B, Zhou L, Zeng C. (-)-Epigallocatechin gallate suppresses proliferation of vascular smooth muscle cells induced by high glucose by inhibition of PKC and ERK1/2 signalings. J Agric Food Chem. 2011 Nov 9;59(21):11483-90. doi: 10.1021/jf2024819. Epub 2011 Oct 14. PMID 21973165